CLINICAL TRIAL: NCT04660084
Title: Impact of Molecular Testing on Improved Diagnosis, Treatment and Management of CAP in Norway: a Pragmatic Randomised Controlled Trial
Brief Title: Impact of Molecular Testing on Improved Diagnosis, Treatment and Management of CAP
Acronym: CAPNOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was stopped earlier than planned after an ad hoc interim analysis
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Drammen sykehus (Other); University of Copenhagen (Other); Rigshospitalet, Denmark (Other); UMC Utrecht (Other); University of Southampton (Other); Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HaukelandUH_31935
Record Dates: First submitted 2020-11-12; First posted 2020-12-09 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2022-03

CONDITIONS: Pneumonia
Keywords: Microbiology; Bacteria and viruses; Rapid diagnosis; Antibiotic resistance; Diagnostic stewardship
MeSH Terms: conditions — Pneumonia; Virus Diseases

STUDY DESIGN:
Intervention Model Description: A pragmatic, parallel-arm, single-blinded, single-centre, randomised controlled superiority trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ultra-rapid molecular point-of-care testing (Other): Extended and more rapid diagnostics on microbiological specimens and an active feedback to treating staff with results.
  Interventions: Diagnostic Test: Ultra-rapid molecular point-of-care testing
- Standard of care (No Intervention): Standard collection of microbiological specimens and standard reply to treating staff.

INTERVENTIONS:
Diagnostic Test: Ultra-rapid molecular point-of-care testing — Ultra-rapid molecular testing (UR-MT) comprises automated detection using the new BioFire® FilmArray® Pneumonia plus platform (Biomérieux). The total turn-around time is <2 hrs.
  The UR-MT is combined with standard of care, comprising:
  Microbiological processing per current standard of care entails culture of respiratory tract samples according to national protocols to detect respiratory bacteria, identified using biochemical methods and/or matrix-assisted laser desorption/ionization time-of-flight (MALDI-TOF MS). Respiratory viruses are identified using real-time PCR (for metapneumovirus, rhinovirus, influenza A, influenza B, parainfluenza 1-3, RSV and SARS-CoV-2). The total turn-around time is up to 48 hrs.
  Other Names: BioFire® FilmArray® Pneumonia plus platform (Biomérieux)
  Arms: Ultra-rapid molecular point-of-care testing

SUMMARY:
Investigators will recruit patients suspected of community-acquired pneumonia at Haukeland University Hospital, Bergen, into a pragmatic randomized controlled trial to assess if provision of ultra-rapid, high-quality accurate molecular diagnostics with direct feedback to the clinician can facilitate pathogen-directed usage of antibiotics, shorten antibiotic exposure and admission time and is safe. Additionally, transcriptional and immune marker profiling of patients will guide appropriate management through a targeted focus on the individual patient's physical capacity, nutritional status and co- morbidities. The pragmatic design of this trial together with broad inclusion criteria and a straightforward intervention would make our results generalisable to other similar centres.

DETAILED DESCRIPTION:
The study is a pragmatic, single-blind, single-centre randomised controlled trial (RCT) where community-acquired pneumonia (CAP) patients will receive standard of care microbiological testing or standard of care microbiological testing and comprehensive ultra-rapid molecular testing (UR-MT).

Investigators will over a 3-year period (2020-2022), consecutively enroll cases of CAP admitted (~900/year) to Haukeland University Hospital (HUS, Bergen). The study will consist of representative patients admitted with CAP and thus, will potentially be generalisable to hospitalised patients with CAP in Norway. As COVID-19 cannot be distinguished clinically from other pneumonias, the study will therefore include patients with suspected CAP, including with COVID-19. Approximately 1500 CAP patients will be screened to achieve a total of 1060 (allowing for a 10% dropout rate) enrolled patients that are randomly assigned to receive standard of care microbiological testing or standard of care testing microbiological and the comprehensive ultra-rapid molecular test (UR-MT).

Inclusion criteria for the study are: adults (aged ≥18 years), with a clinical diagnosis of CAP (presence of at least two clinical criteria [new/worsening cough, new/worsening expectoration of sputum, haemoptysis, new/worsening dyspnoea, pleuritic chest pain, fever, or abnormalities on chest auscultation or percussion] or one clinical criterion and radiological evidence of CAP), requiring hospitalisation to a non-ICU ward, and with a capacity to give informed written consent or consent provided by the patient's legally authorized representative.

Exclusion criteria include: lung tumour, cystic fibrosis, a palliative approach, patients who decline to provide respiratory tract specimens, severe immunodeficiency, and hospitalization for two or more days in the last 14 days.

Based on clinical evaluation and data of admission, patients will be triaged for severity according to current risk assessment guidelines, as well as the CRB-65 score for the assessment of severity of pneumonia. Randomization of CAP patients to the two treatment arms (1:1) will be performed in blocks of size 4, 6, or, 8, occurring in random order, to ensure approximately equal allocation over the year.

The prescribed empirical therapy for each patient will be compared with what antimicrobial(s) would have been appropriate for pathogen-directed therapy, based on the UR-MT result. Appropriate pathogen-directed therapy will be determined using national guidelines recommended by the Norwegian directorate of health

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥18 years),
* Clinical diagnosis of CAP (presence of at least two clinical criteria [new/worsening cough, new/worsening expectoration of sputum, haemoptysis, new/worsening dyspnoea, pleuritic chest pain, fever, or abnormalities on chest auscultation or percussion] or one clinical criterion and radiological evidence of CAP)
* Requiring hospitalisation to a non-ICU ward
* Capacity to give informed written consent or consent provided by the patient's legally authorized representative.

Exclusion Criteria:

* Pulmonary embolism
* Lung tumor
* Cystic fibrosis
* Palliative approach
* Patients who decline to provide respiratory tract specimens
* Severe immunodeficiency
* Hospitalization for two or more days in the last 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
The provision of pathogen-directed treatment based on a microbiological test result deemed as clinically relevant within 48 hours of receipt of respiratory samples. | "Up to 72 hours"
  Binary outcome: yes: it was provided/no: it was not provided
Time in hours from receipt of respiratory specimens to receiving pathogen-directed treatment | "Up to 72 hours"
  Quantitative outcome (measured in hours): time from receipt of respiratory specimens to provision of pathogen-directed treatment based on a microbiological test result deemed as clinically relevant or an elapse of 48 hours, whichever event came first.

SECONDARY OUTCOMES:
Duration of antibiotic use in days | "Up to 4 weeks"
  Duration of antibiotic use in days
Proportion of patients receiving narrow-spectrum antibiotics within 48 hours from study inclusion | "Up to 4 weeks"
  Proportion of patients receiving narrow-spectrum antibiotics within 48 hours from study inclusion
Proportion of patients receiving a single dose of antibiotics | "Up to 1 week"
  Proportion of patients receiving a single dose of antibiotics
Proportion of patients receiving ≤48 h of antibiotics | "Up to 1 week"
  Proportion of patients receiving ≤48 h of antibiotics
Proportion of patients receiving intravenous antibiotics | "Up to 1 week"
  Proportion of patients receiving intravenous antibiotics
Duration of intravenous antibiotics in days | "Up to 4 weeks"
  Duration of intravenous antibiotics in days
Proportion of cases where the UR-MT results were used to guide treatment | "Up to 1 week"
  Proportion of cases where the UR-MT results were used to guide treatment
Time in days to isolation or de-isolation | "Up to 2 weeks"
  Time in days to isolation or de-isolation
Duration of "door-to-needle time" in hours | "Up to 1 week"
  Duration of "door-to-needle time" in hours
Length of hospital stay in days | "Up to 3 months"
  Length of hospital stay in days
Proportion of 30-day readmission | "Up to 30 days from discharge"
  Proportion of 30-day readmission
Proportion of 30- and 90-day and 1- and 5 year mortality | "Up to 1 month, 3 months, 1 and 5 years, from admission"
  Proportion of 30- and 90-day and 1- and 5 year mortality

CONTACTS AND LOCATIONS:
Overall Officials: Harleen Grewal, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saghaug CS, Markussen DL, Knoop ST, Holvik BC, Serigstad S, Ulvestad E, Ritz C, Jenum S, Grewal HMS. Diagnostic accuracy of a host response test in suspected community-Acquired pneumonia during the COVID-19 era. Int J Infect Dis. 2025 Nov;160:108045. doi: 10.1016/j.ijid.2025.108045. Epub 2025 Sep 2. PMID 40907740
- [Derived] Markussen DL, Wathne JS, Ritz C, van Werkhoven CH, Serigstad S, Bjorneklett RO, Ulvestad E, Knoop ST, Jenum S, Grewal HMS. Determinants of non-adherence to antibiotic treatment guidelines in hospitalized adults with suspected community-acquired pneumonia: a prospective study. Antimicrob Resist Infect Control. 2024 Nov 23;13(1):140. doi: 10.1186/s13756-024-01494-2. PMID 39580437
- [Derived] Markussen DL, Serigstad S, Ritz C, Knoop ST, Ebbesen MH, Faurholt-Jepsen D, Heggelund L, van Werkhoven CH, Clark TW, Bjorneklett RO, Kommedal O, Ulvestad E, Grewal HMS. Diagnostic Stewardship in Community-Acquired Pneumonia With Syndromic Molecular Testing: A Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e240830. doi: 10.1001/jamanetworkopen.2024.0830. PMID 38446481
- [Derived] Markussen DL, Ebbesen M, Serigstad S, Knoop ST, Ritz C, Bjorneklett R, Kommedal O, Jenum S, Ulvestad E, Grewal HMS. The diagnostic utility of microscopic quality assessment of sputum samples in the era of rapid syndromic PCR testing. Microbiol Spectr. 2023 Sep 29;11(5):e0300223. doi: 10.1128/spectrum.03002-23. Online ahead of print. PMID 37772853
- [Derived] Serigstad S, Knoop ST, Markussen DL, Ulvestad E, Bjorneklett RO, Ebbesen MH, Kommedal O, Grewal HMS. Diagnostic utility of oropharyngeal swabs as an alternative to lower respiratory tract samples for PCR-based syndromic testing in patients with community-acquired pneumonia. J Clin Microbiol. 2023 Sep 21;61(9):e0050523. doi: 10.1128/jcm.00505-23. Epub 2023 Aug 16. PMID 37585220
- [Derived] Serigstad S, Ritz C, Faurholt-Jepsen D, Markussen D, Ebbesen MH, Kommedal O, Bjorneklett RO, Heggelund L, Clark TW, van Werkhoven CH, Knoop ST, Ulvestad E, Grewal HMS; CAPNOR study group. Impact of rapid molecular testing on diagnosis, treatment and management of community-acquired pneumonia in Norway: a pragmatic randomised controlled trial (CAPNOR). Trials. 2022 Aug 1;23(1):622. doi: 10.1186/s13063-022-06467-7. PMID 35915452